CLINICAL TRIAL: NCT04629638
Title: Maternal Attachment and Depression Anxiety Score Evaluation in COVID-19 Positive Pregnant Women
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: maternalattachmentcovid
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Depression, Anxiety; Pregnancy Related
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid -19 positive pregnant women: Maternal attachment, Edinburgh depression scoring, and postpartum anxiety scale are evaluated in 250 covid-positive pregnant women in the 3rd month after birth.
  Interventions: Other: Maternal attachment, Edinburgh depression scoring and postpartum anxiety scale scores
- covid -19 negative pregnant women: Maternal attachment, Edinburgh depression scoring, and postpartum anxiety scale are evaluated in 250 covid-negative pregnant women in the 3rd month after birth.
  Interventions: Other: Maternal attachment, Edinburgh depression scoring and postpartum anxiety scale scores

INTERVENTIONS:
Other: Maternal attachment, Edinburgh depression scoring and postpartum anxiety scale scores — The results will be compared with the results of covid-negative pregnant women who gave birth in the same period.

SUMMARY:
Maternal attachment, Edinburgh depression scoring, and postpartum anxiety scale are evaluated in patients with covid-positive pregnancies in the 3rd month after birth.

DETAILED DESCRIPTION:
Maternal attachment, Edinburgh depression scoring and postpartum anxiety scale are evaluated in 250 covid-positive pregnant women in the 3rd month after birth. The results will be compared with the results of covid-negative pregnant women who gave birth in the same period.

ELIGIBILITY:
Inclusion Criteria:

* covid -19 positive and negative pregnant women
* have no psychiatric illness
* not using antidepressants or antipsychotic drugs

Exclusion Criteria:

* women with psychiatric illness
* using antidepressants or antipsychotic drugs
* not pregnant
* adolescent pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Maternal attachment, edinburgh depression score and postpartum anxiety scale scores of 250 covid-19 positive pregnant women between the ages of 18-45 and 250 covid-negative pregnant women are compared.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Maternal attachment in SARS- cov2 positive and negative pregnant women | 3 months
  Maternal attachment scores evaluated in 250 covid-positive pregnant women in the 3rd month after birth. The results will be compared with the results of covid-negative pregnant women who gave birth in the same period. High scores from the scale indicate high maternal attachment.
Edinburgh depression scores in in SARS- cov2 positive and negative pregnant women | 3 months
  Edinburgh depression scores evaluated in 250 covid-positive pregnant women in the 3rd month after birth. The results will be compared with the results of covid-negative pregnant women who gave birth in the same period. All questions are scored between 0 and 3 and the highest possible score on the scale is 30. and shows advanced depression.
Postpartum anxiety scale scores in in SARS- cov2 positive and negative pregnant women | 3 months
  Postpartum anxiety scale scores evaluated in 250 covid-positive pregnant women in the 3rd month after birth. The results will be compared with the results of covid-negative pregnant women who gave birth in the same period. It can be said that the postpartum anxiety levels of those who score 73 and below on the scale are low, those who score between 74 and 100 are medium, and those who score 101 and above are high.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No